CLINICAL TRIAL: NCT07206043
Title: Single-Center, Randomized, Cohort, Single-Blind, Comparative Clinical Study to Evaluate the Pharmacokinetics, Safety, and Immunogenicity of RPH-104 in a New 80 mg/mL Dosage Form Following Single Subcutaneous and Intravenous Administration at Doses of 80 mg, 160 mg, and 320 mg in Healthy Volunteers
Brief Title: Pharmacokinetics, Safety and Immunogenicity of RPH-104 at a New Dosage and Different Doses Via Single Subcutaneous and Intravenous Administration in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: R-Pharm International, LLC (Industry)
Collaborators: LLC "Exacte Labs" (Unknown); JSC "R-Pharm", Russia (R-Pharm Group) (Unknown)
Responsible Party: Sponsor
Organization: R-Pharm (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CL04018366
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: subcutaneous; intravenous; Anti-IL1; Anti-IL1 beta; RPH-104

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Cohort A: RPH-104, intravenous administration 80 mg (Experimental): Subjects received RPH-104 Intravenously once as a 60-minute infusion at a dosage of 40 mg/mL, at a dose of 80 mg. The volume of the infusion solution was 100 ± 8 mL
  Interventions: Biological: RPH-104 80 mg
- Cohort A: RPH-104, intravenous administration 160 mg (Experimental): Subjects received RPH-104 Intravenously once as a 60-minute infusion at a dosage of 40 mg/mL, at a dose of 160 mg. The volume of the infusion solution was 100 ± 8 mL
  Interventions: Biological: RPH-104 160 mg
- Cohort A: RPH-104, intravenous administration 320 mg (Experimental): Subjects received RPH-104 Intravenously once as a 60-minute infusion at a dosage of 40 mg/mL, at a dose of 320 mg. The volume of the infusion solution was 100 ± 8 mL
  Interventions: Biological: RPH-104 320 mg
- Cohort B: RPH-104, subcutaneous administration 320 mg (Experimental): Subjects received a single subcutaneous injection of either RPH-104 at a dosage of 80 mg/mL, at a dose of 320 mg (2 injections of 2 mL), or a placebo (2 injections of 2 mL)
  Interventions: Biological: RPH-104 320 mg
- Cohort B: Placebo (Placebo Comparator): Placebo Comparator, Placebo
  Interventions: Drug: Placebo
- Cohort C: RPH-104, subcutaneous administration 80 mg (40 mg/mL) (Experimental): Subjects received a single subcutaneous injection of either RPH-104 at a dosage of 40 mg/mL, at a dose of 80 mg (1 injection of 2 mL)
  Interventions: Biological: RPH-104 80 mg
- Cohort C: RPH-104, subcutaneous administration 80 mg (80 mg/mL) (Experimental): Subjects received a single subcutaneous injection RPH-104 at a dosage of 80 mg/mL, at a dose of 80 mg (1 injection of 1 mL)
  Interventions: Biological: RPH-104 80 mg

INTERVENTIONS:
Biological: RPH-104 80 mg — solution for intravenous injection, 40 mg/mL
  Other Names: goflikicept
  Arms: Cohort A: RPH-104, intravenous administration 80 mg
Biological: RPH-104 160 mg — solution for intravenous injection, 40 mg/mL
  Other Names: goflikicept
  Arms: Cohort A: RPH-104, intravenous administration 160 mg
Biological: RPH-104 320 mg — solution for intravenous injection, 40 mg/mL
  Other Names: goflikicept
  Arms: Cohort A: RPH-104, intravenous administration 320 mg
Biological: RPH-104 320 mg — solution for subcutaneous injection, 80 mg/mL
  Other Names: goflikicept
  Arms: Cohort B: RPH-104, subcutaneous administration 320 mg
Biological: RPH-104 80 mg — solution for subcutaneous injection, 40 mg/mL
  Other Names: goflikicept
  Arms: Cohort C: RPH-104, subcutaneous administration 80 mg (40 mg/mL)
Biological: RPH-104 80 mg — solution for subcutaneous injection, 80 mg/mL
  Other Names: goflikicept
  Arms: Cohort C: RPH-104, subcutaneous administration 80 mg (80 mg/mL)
Drug: Placebo — 0.9% Sodium Chloride solution for Injection
  Arms: Cohort B: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, immunogenicity and pharmacokinetics of RPH-104 after single intravenous and subcutaneous administration to healthy volunteers at different doses

DETAILED DESCRIPTION:
This clinical study is a single-center, simple-blind, randomized, comparative phase I clinical study conducted in 3 parallel cohorts:

In cohort A, a simple blind design is proposed with a single intravenous administration of the study drug at 3 increasing doses (N = 30, 10 volunteers per dose group): 80 mg, 160 mg, 320 mg

In cohort B, a simple blind design is proposed with a single subcutaneous administration of the study drug (80 mg/mL; 320 mg) compared to placebo (N = 20, 10 volunteers per drug and placebo group)

In cohort C, a simple blind design is proposed with a single subcutaneous administration of the study drug in two dosages (40 mg/mL and 80 mg/mL) in one dose (80 mg) to confirm the equivalence of these dosages (N = 80, 40 volunteers in each group)

The study will include the following periods:

1. Screening period: days -6 to -1 (before randomization and inclusion in the study)
2. Randomization: day 0
3. Main study period:days 1 to 50 (± 1)

   The main period includes a single hospitalization of volunteers for at least 24 hours, as well as 9 outpatient visits in cohort A and 14 outpatient visits in cohorts B and C. It includes procedures related to the administration of the study drug, monitoring the study participant, and taking blood samples to measure the concentration of goflikicept, as well as a safety and immunogenicity panel
4. Safety monitoring period: days 51 - 61 (± 3). On day 61, a phone call will be made to collect information about safety

In order to monitor safety during the main sudy period, the following procedures will be carried out:

* In Cohort A, vital signs vital signs will be measured before drug administration and 15 min, 1 h, 2 h, 4 h, 12 h and 24 h after drug administration on days 3-50; physical examination will be performed on days 2, 6, 16, 30, 40, 50; electrocardiography (ECG) on days 3, 23, 50 day; assessment of hypersensitivity reactions to the drug in 2 h, 12 h, 24 h after the start of drug administration and on day 3; clinical blood test, biochemical blood test on 3, 6, 16, 23, 50 day; coagulogram on 3, 16, 50 day; general urinalysis on 6, 16, 23, 50 day.
* In Cohort B and C, vital signs vital signs will be measured before drug administration and in 2 h, 12 h and 24 h after drug administration on days 3-50; physical examination will be performed on days 2, 6, 16, 30, 40, 50; ECG on days 5, 23, 50 day; assessment of hypersensitivity reactions to the drug in 2 h, 12 h, 24 h after the start of drug administration and on day 3; clinical blood test, biochemical blood test on 5, 9, 16, 30, 50 day; coagulogram on 5, 16, 50 day; general urinalysis on 5, 16, 30, 50 day
* Women with preserved reproductive potential will additionally undergo blood analysis for hCG during screening, followed by a urine pregnancy test the day before the administration of RPH-104 (Day 0) and on Day 50

To assess the pharmacokinetics of RPH-104, volunteers will undergo periodic blood sampling (at a total of 18 points during the study for cohort A, and at 18 points for cohorts B and C)

* In cohort A, blood samples for the evaluation of RPH-104 pharmacokinetics will be taken before the infusion of RPH-104 on Day 1 (< 60 min before infusion ) and in 30 min, 1 h (immediately after the end of the infusion), 1 h and 30 min, 2 h, 4 h, 8 h, 12 h, 24 h, 48 h, 72 h, 120 h, 192 h, 360 h, 528 h, 696 h, 936 h and 1176 h after the first administration of the drug (since the start of infusion)
* In cohort B and C, blood samples for the evaluation of RPH-104 pharmacokinetics will be taken before the infusion of RPH-104 on Day 1 (< 60 min before infusion ) and in 4 h, 12 h, 24 h, 48 h, 72 h, 84 h, 96 h, 108 h, 144 h,120 h, 192 h, 264 h, 360 h, 528 h, 696 h, 936 h and 1176 h after the first administration of the drug (since the start of infusion)

To assess the immunogenicity of RPH-104, volunteers will undergo periodic blood sampling to determine the concentration of binding and neutralizing antibodies (at a total of 5 points in the study in all cohorts)

* In cohort A, blood sampling for immunogenicity testing is performed before the drug is administered (≤60 min before administration) and then in 360 h (day 16) (± 120 min), 696 h (day 30) (±24 h), 936 h (day 40) (±24 h), 1176 h (day 50) (±24 h) after administration of the drug. When binding antibodies are detected, their neutralizing activity (NAT) will additionally be determined
* In cohort B and C, blood sampling for immunogenicity testing is performed before the drug is administered (≤60 min before administration) and then in 360 h (day 16) (± 120 min), 696 h (day 30) (±24 h), 936 h (day 40) (±24 h), 1176 h (day 50) (±24 h) after administration of the drug. When binding antibodies are detected, their neutralizing activity (NAT) will additionally be determined

ELIGIBILITY:
Volunteers had to meet all the following inclusion criteria:

1. Signed and dated Informed Consent Form in duplicate
2. Males and females aged 18-45 years inclusive
3. Body mass index:

   * Cohorts A and B: normal range (18.5-29.9 kg/m²)
   * Cohort C: normal range (18.5-29.9 kg/m²), body mass ≥55 and ≤100 kg
4. Verified "healthy" diagnosis per standard clinical, laboratory, and instrumental examinations:

   1. Normal results for complete blood count, blood chemistry, coagulation tests, urinalysis, and ECG per center standards (screening tests performed ≤7 days before enrollment)
   2. Normal vital signs: SBP 90-129 mmHg, DBP 60-85 mmHg, pulse 60-100 bpm, body temperature 36.1-37.0℃, respiratory rate 12-20 breaths/min
   3. No tuberculosis (active, latent, or history) or other chronic infections/inflammatory diseases
   4. Satisfactory health status (per volunteer's opinion) for 30 days prior to consent
   5. "Normal" result for physical examination by investigator's judgment at screening
5. Agreement to abstain from alcohol for 72 hours pre-dose until final PK blood sampling
6. Willingness to comply with protocol procedures per investigator's judgment
7. Agreement (by volunteers and their partners of reproductive potential for male volunteers) to abstain from heterosexual intercourse or use highly effective contraception from consent until 3 months post-goflikicept administration
8. For female volunteers: willingness to consent to pregnancy outcome data collection and provide obstetric/pediatric clinic contacts if pregnancy occurs post-dosing

Subjects were withdrawn from further participation in the study in the following cases:

1. Detection, after inclusion of the subject in the study, of non-compliance with the inclusion criteria or presence, at the time of inclusion, of compliance with the exclusion criteria (as decided by LLC "R-Pharm International", including retrospective analysis of information entered into the eCRF database)
2. If the subject withdraws their consent to participate in the study
3. If AEs or SAEs, laboratory abnormalities, or concomitant diseases are identified in the subject, which, in the opinion of the investigator or the Sponsor, make continued participation impossible or dangerous, or not in the best interest of the subject's welfare and safety
4. In case of subject non-compliance (in this case, exclusion of the subject must be agreed upon with representatives of LLC "R-Pharm International", see Section 6.3 of the Clinical Study Protocol), or in the case of systematic major deviations in the timing of scheduled visits (more than 3 deviations from scheduled visit dates). For Cohort C: in case of missing any of Visits 09, missing two consecutive Visits 1015, or missing any 3 visits during the study
5. If the study is terminated by decision of LLC "R-Pharm International", local ethics committees, or regulatory authorities
6. In case of use of drugs prohibited by the Protocol
7. If restrictions for study subjects are violated (in this case, exclusion of the subject must be agreed upon with representatives of LLC "R-Pharm International", see Section 6.2.3 of the Clinical Study Protocol "Other restrictions for study subjects")
8. If there is suspicion of concurrent participation in another clinical study, including indirect laboratory evidence
9. If the result of a test for alcohol, narcotic, or psychotropic substances is positive before administration of the study drug
10. If SARS-CoV-2 is detected via PCR test or rapid antigen test prior to administration of the study drug
11. If other reasons arise during the study that prevent the study from being conducted according to the protocol
12. In the event of the subject's death
13. For female subjects a positive pregnancy test (test strip), performed at the center prior to administration of the study drug
14. In case of missed blood sample collections (applicable only for Cohort C)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
The area under the plasma drug concentration-time curve (AUC) of RPH-104 from the moment of administration to infinity after a single injection of RPH-104 | Up to day 61 ± 3
  The area under the plasma drug concentration-time curve (AUC) of RPH-104 from the moment of administration to infinity after a single injection of RPH-104 (AUC(0-∞))
The maximum concentration of RPH-104 in the blood serum after a single injection of RPH-104 | Up to day 61 ± 3
  The maximum concentration of RPH-104 in the blood serum after a single injection of RPH-104 (Cmax).
Percentage of volunteers (%) with AEs and SAEs | Up to day 61 ± 3
  Percentage of volunteers (%) with AEs and SAEs
Percentage of volunteers (%) with AEs ≥ Grade 3 according to CTCAE 5.0 | Up to day 61 ± 3
  Percentage of volunteers (%) with AEs ≥ Grade 3 according to CTCAE 5.0
Percentage of volunteers (%) with ADRs and serious ADRs | Up to day 61 ± 3
  Percentage of volunteers (%) with ADRs and serious ADRs
Percentage of volunteers (%) with ADRs ≥ Grade 3 according to CTCAE 5.0 | Up to day 61 ± 3
  Percentage of volunteers (%) with ADRs ≥ Grade 3 according to CTCAE 5.0
Percentage of volunteers (%), who prematurely discontinued participation in the study due to AE/SAE and ADR/serious ADR | Up to day 61 ± 3
  Percentage of volunteers (%), who prematurely discontinued participation in the study due to AE/SAE and ADR/serious ADR
Percentage of volunteers (%) with AEs of special interest | Up to day 61 ± 3
  AEs of special interests include allergic and anaphylactic reactions, injection site reactions, infections, increased blood lipid levels, increased liver enzyme levels, drug-induced liver injury, neutropenia
Percentage of volunteers (%), who developed binding antibodies to RPH-104 | Up to day 61 ± 3
  Percentage of volunteers (%), who developed binding antibodies to RPH-104
Percentage of volunteers (%), who developed neutralizing antibodies to RPH-104 | Up to day 61 ± 3
  Percentage of volunteers (%), who developed neutralizing antibodies to RPH-104

SECONDARY OUTCOMES:
The area under the plasma drug concentration-time curve (AUC) of RPH-104 from the moment of administration to the last time point of sampling | Up to day 50 ± 1
  The area under the plasma drug concentration-time curve (AUC) of RPH-104 from the moment of administration to the last time point of sampling (AUC(0-1176))
The time to reach the maximum concentration of RPH-104 after a single injection | Up to day 50 ± 1
  The time to reach the maximum concentration of RPH-104 after a single injection (Tmax)
Apparent total clearance of RPH-104 after a single administration | Up to day 50 ± 1
  Apparent total clearance of RPH-104 after a single administration (Cl/F)
The half-life of RPH-104 after a single administration | Up to day 50 ± 1
  The half-life of RPH-104 after a single administration (T1/2)
The apparent volume of distribution of RPH-104 after a single administration | Up to day 50 ± 1
  The apparent volume of distribution of RPH-104 after a single administration (Vd/F)
The elimination constant of RPH-104 after a single administration | Up to day 50 ± 1
  The elimination constant of RPH-104 after a single administration (λz)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — R-Pharm
Locations (1):
- Llc "Research Lab", Moscow, Russia